CLINICAL TRIAL: NCT03283644
Title: Obesity-related Inflammation in Patients Prior to and After Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: University of Birmingham (Other)
Collaborators: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: ERN_13-0355
Record Dates: First submitted 2017-02-08; First posted 2017-09-14 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2017-02

CONDITIONS: Obesity; Morbid Obesity
Keywords: gastric bypass; Obesity; Morbid obesity; Matched Healthy Controls
MeSH Terms: conditions — Obesity; Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with a BMI over 40: Participants were aged between 27-65 years, BMI >40 , Co-Morbidities associated with obesity including sleep apnoea, hypertension, depression, hypercholesterolaemia and type 2 diabetes, Undergoing Gastric Band surgery
- Lean, healthy individuals: Participants were aged between 27-65 years, BMI<28 , Systemically healthy, taking no prescribed medication

SUMMARY:
This study investigates the chronic long-term health condition of obesity and its effect on neutrophil function and the inflammatory response

DETAILED DESCRIPTION:
Inflammation is a central component of the immune response. In its acute form it aids the transition from disease to health via the activation of numerous immune cells, enabling them to reach the site of infection/injury and orchestrate themselves to combat pathogens, facilitating resolution and repair to restore the host to health. However, chronic inflammation is deleterious to the host and differs from the "classical" acute inflammatory process in that the inflammation is not necessarily so readily obvious and is not self-limiting; rather, the immune system is in a constant state of low-grade activation and when challenged by pathogenic or sterile injury the response is heightened, resulting in prolonged tissue damage and a failure of efficient resolution mechanisms.

Neutrophils are important mediators of acquired innate immune responses but may also contribute to the pathogenesis of chronic inflammatory diseases. Neutrophils are heavily involved in antimicrobial defence; their primary role is the localisation and elimination of pathogenic microorganisms. This, combined with their relatively short lifespan, has resulted in a traditional view of them as limited "kamikaze" cells. However, as detailed here, neutrophils have been shown to act with complexity and sophistication, orchestrating the immune/inflammatory response but also inadvertently contributing to tissue damage in different disease states. This study investigates the chronic long-term health condition of obesity and its effect on neutrophil function and the inflammatory response

ELIGIBILITY:
Inclusion Criteria for Bariatric participants:

* BMI >40
* Undergoing Gastric Band surgery

Exclusion Bariatric Participants Criteria:

* Undergoing alternative weight loss surgery
* BMI<40
* Smoking
* Pregnancy

Exclusion criteria for the controls

* BMI over 27
* pregnancy
* smoking
* evidence of systemic disease
* use of medications/vitamin supplements.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two study populations: Healthy control defined as systemically healthy and not taking medication or supplements with a BMI less than 27; Bariatric participants who fit the inclusion and exclusion criteria, but may also present with co-morbidities associated with obesity.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-08-28 (Actual); Study Completion 2016-10-28 (Actual)

PRIMARY OUTCOMES:
Biochemical Markers associated with Inflamation | OCT 2016
  (IL-8, IL-1, ROS, Production of NETS)

IPD SHARING:
Plan to Share IPD: No